CLINICAL TRIAL: NCT07102680
Title: A RANDOMIZED PLACEBO CONTROLLED TRIAL OF L MAX IN HEALTHY ADULT ATHLETES
Brief Title: A Randomized, Placebo Controlled Trial of L Max in Healthy Adult Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Climatic, Inc. (Industry)
Collaborators: People Science (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CHI-A2-001
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Healthy Normal Athletes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L Max Arm (Active Comparator): Participants will complete up to a ten week study consisting of screening period, pre-study preparation period, baseline period, a 4-week product use period. Screening assessments, baseline questions, participant reported outcome surveys, exercise, health, and dosing logs, and adverse event reporting will be collected. Participants will have the option of participating in an end of study interview. This study will be conducted remotely and will use a web-based data collection platform, Consumer Health Learning and Organizing Ecosystem (Chloe), by People Science where participants will complete study assessments using the Chloe app during the course of the study. Participants will receive the study product during the pre-study preparation period. Demographic and limited medical history data will be collected for the study.
  Interventions: Other: L Max
- Placebo Arm (Placebo Comparator): Participants will complete up to a ten week study consisting of screening period, pre-study preparation period, baseline period, a 4-week product use period. Screening assessments, baseline questions, participant reported outcome surveys, exercise, health, and dosing logs, and adverse event reporting will be collected. Participants will have the option of participating in an end of study interview. This study will be conducted remotely and will use a web-based data collection platform, Consumer Health Learning and Organizing Ecosystem (Chloe), by People Science where participants will complete study assessments using the Chloe app during the course of the study. Participants will receive the study product during the pre-study preparation period. Demographic and limited medical history data will be collected for the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: L Max — L Max proprietary formulation
  Arms: L Max Arm
Other: Placebo — Lactohale 300
  Arms: Placebo Arm

SUMMARY:
The goal of this study is to evaluate the lung-cleansing effects of L Max by measuring changes in Participant Reported Outcome (PRO) Scores and athletic performance. Researchers will compare the results of participants who take L Max and participants who take placebo (a look-alike substance that contains no active ingredient).

Participants will:

1. Wear an Oura Ring continuously throughout the study
2. Perform spirometry (a measurement of your lung health) daily
3. Fill out short daily exercise and health logs
4. Perform three timed athletic performance tests over the course of the study and record the results
5. Fill out Participant Reported Outcomes Surveys three times over the course of the study
6. Fill out study product surveys twice over the course of the study
7. Participate in an optional exit survey at the end of the study

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 60 years
2. US-based
3. Committed endurance athlete with cycling, triathlon or running focus
4. Achieves three or more Zone 3+ sessions/week
5. Tracks power and time during training
6. Able to use Oura, spirometry, and training apps
7. Routinely feels pulmonary system/breathing limits athletic performance
8. If diagnosed with exercise induce asthma, able to use inhaler only as rescue and not preventatively.
9. Women of childbearing potential (WOCBP) must agree to use highly effective contraception starting at least 14 days prior to the first dose of L Max or placebo, throughout the study period, and for at least 30 days after the last dose of study product.

   Highly effective methods include the following: abstinence, oral contraceptives, contraceptive injections, intrauterine device, double barrier method (Diaphragm or condom + spermicidal cream) contraceptive patch, or male partner sterilization. Women who are postmenopausal (at least 12 months of spontaneous amenorrhea without an alternative medical cause) or surgically sterile (e.g. hysterectomy, salpingectomy, bilateral oophorectomy, or bilateral tubal ligation) are not considered of childbearing potential.
10. Willing to practice a reliable method of contraception for the duration of the study
11. In good general health at the time of screening (Investigator discretion).
12. Able to read and understand English
13. Able to read, understand, and provide informed consent
14. Able to use a personal smartphone device and download Chloe by PeopleScience, Oura, and MIR Spirobank
15. Able to receive shipment of the product at an address within the United States
16. Able to complete study assessments over the course of up to 6 weeks.

Exclusion Criteria:

1. Do not have a personal smartphone, internet access, or are unwilling to download Chloe, Oura, or MIR Spirobank apps
2. Daily/preventative inhaler use
3. Injury, illness, or poor training compliance in the previous 6 months
4. History of COPD, long COVID, fibromyalgia, chronic fatigue syndrome, Lyme disease, or major cardiac or respiratory conditions
5. Lack of access to indoor trainer with power meter
6. High alcohol use or ongoing recreational drug/tobacco use
7. Pregnant, planning to become pregnant during the study, or lactating
8. Use of medications to treat hypertension (high blood pressure) including diuretics, Angiotensin Converting Enzyme inhibitors, Angiotensin II Receptor Blockers, calcium channel blockers, beta blockers, alpha blockers, and other classes used for blood pressure control
9. Any underlying medical conditions or comorbidities that may confound the assessment or the evaluation of the study outcomes.
10. Have a significant illness, disease, or condition which, in the opinion of the principal investigator, may impact their ability to participate in the study or impact the study outcomes.
11. Known hypersensitivity or previous allergic reaction to sodium bicarbonate, citrate, theobromine, arginine, forskolin, maltodextrin, modified food starch, or lactose
12. Are unlikely for any reason to be able to comply with the trial or are considered unsuited for participation in the study by the Principal Investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Composite PRO Score | From baseline to the end of treatment at 42 days
  Change from baseline between placebo and study groups of the Composite PRO score. Composite PRO is comprised of 4 questions related to the participant's experience during Zone 3+ workouts. Score ranges from 9 to 45, higher scores indicating better outcome.
Change from baseline in Composite PRO Question #1 | From baseline to end of treatment at Day 42
  Change from baseline between placebo and study groups on question #1: Over the past two weeks, how would you rate any changes in your breathing, congestion, or overall lung health during high-intensity workouts (Zone 3+) compared to your normal baseline? Score ranges from 1 to 5, higher score indicating better outcome.
Change from baseline in Composite PRO Question #2 | From baseline to end of treatment at Day 42
  Change from baseline between placebo and study groups on question #2: Over the past two weeks, how would you rate your ease of breathing during high-intensity workouts (Zone 3+)? Score ranges from 1 to 5, higher score indicating better outcome.
Change from baseline in Composite PRO Question #3 | From baseline to end of treatment at Day 42
  Change from baseline between placebo and study groups on question #3: Over the past two weeks, how often do you experience the following during high-intensity workouts (Zone 3+): Shortness of breath, Chest tightness, Wheezing, Coughing, Fatigue or difficulty maintaining intensity, Phlegm or mucus buildup? Scores range from 1 to 5 for each element, higher score indicating better outcome.
Change from baseline in Composite PRO Question #4 | From baseline to end of treatment at Day 42
  Change from baseline between placebo and study groups on question #4: Over the last two weeks, how would you rate your ability to push yourself during high-intensity workouts (Zone 3+)? Score ranges from 1 to 5, higher number indicating better outcome.

SECONDARY OUTCOMES:
Percent change from baseline in timed performance test completion time | From baseline to end of treatment at Day 42
  Percent change from baseline between placebo and study groups on a timed performance test. The timed performance test will be either a 5k run or 5 mi cycle on an indoor trainer. Participants will focus on all-out effort and will record the time it takes to complete the performance test. The performance test will be completed at baseline and at 2 weeks and 4 weeks of study participation. A faster performance time will indicate improvement.
Percent change from baseline in power output during timed performance test | From baseline to end of treatment at Day 42
  Percent change from baseline between placebo and study groups on a timed performance test. The timed performance test will be either a 5k run or 5 mi cycle on an indoor trainer. Participants will focus on all-out effort and will record the their power output during the performance test. The performance test will be completed at baseline and at 2 weeks and 4 weeks of study participation. A faster performance time will indicate improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Craft Principal Investigator, M.D., Principal Investigator — People Science
Locations (1):
- People Science, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
The data are part of ongoing research and will not be available for sharing due to potential publication and/or intellectual property considerations.